CLINICAL TRIAL: NCT00277394
Title: Safety Profile of Innohep Versus Subcutaneous Unfractionated Heparin in Elderly Patients With Impaired Renal Function Treated for Acute Deep Vein Thrombosis
Brief Title: Innohep® in Elderly Patients With Impaired Renal Function Treated for Acute Deep Vein Thrombosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN 0401 INT
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2019-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Acute, symptomatic and objectively confirmed DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — Tinzaparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- innohep® (Experimental): innohep® 175 anti-Xa IU/kg once daily
  Interventions: Drug: innohep®
- Heparin (Active Comparator): Heparin 50 IU /kg followed by a total dose of 400 to 600 IU/kg/day divided into two SC injections daily.
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: innohep® — 175 anti-Xa IU/kg administered subcutaneously (SC) once daily
  Arms: innohep®
Drug: Heparin — Heparin 50 IU /kg followed by a total dose of 400 to 600 IU/kg/day divided into two SC injections daily.
  Arms: Heparin

SUMMARY:
The objective of the study is to compare the safety of innohep® and Unfractionated Heparin (UFH) in terms of clinically relevant bleedings in elderly patients with impaired renal function for initial treatment of acute Deep Venous Thrombosis (DVT).

The primary response criterion is the percentage of patients with clinically relevant bleeding events prior to day 90 +/- 5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic and objectively confirmed Venous Thromboembolism (VTE) (lower limb deep venous thrombosis (DVT) or pulmonary embolus (PE)) with mandatory presences of objectively confirmed and treatment requiring DVT, i.e. symptomatic and objectively confirmed distal DVT or objectively confirmed, symptomatic or asymptomatic proximal DVT (confirmation of DVT should be performed by ultrasonography or venography within 48 hous prior to randomisation)
* Patients with an indication for DVT treatment with SC Low Molecular Weight Heparin (LMWH) or Unfractionated Heparin (UFH) followed by Oral Anticoagulant (OAC) for at least 90 days
* Hospitalized patients who, during SC anticoagulant treatment, will be followed, as specified in the protocol, on a daily basis either in the hospital or in an out-patient setting
* Patients at or above 75 years with a creatinine clearance less than or equal to 60 mL/min calculated according to the Cockcroft-Gault formula
* Patients at or above 70 years with a creatinine clearance less than or equal to 30 mL/min calculated according to the Cockcroft-Gault formula

Exclusion Criteria:

* Patients receiving high dose (i.e. equivalent to a dose recommended for treatment of DVT) of UFH or LMWH or thrombolytic agents within the last 4 weeks except for UFH/LMWH during the last 36 hours prior to randomisation
* Patients on oral anticoagulant treatment (vitamin K-antagonists) at or within last 1 week prior to randomisation
* Patients with a symptomatic venous thromboembolism (VTE) requiring thrombolytic therapy or invasive intervention
* End stage renal disease patients requiring dialysis
* Surgery within 2 weeks prior to randomisation or planned surgery, epidural anaesthesia and/or spinal anaesthesia during the SC anticoagulant treatment period
* Planned use of acetylsalicylic acid in doses above 300 mg/day, NSAID or Dextran 40 at randomisation and during the SC anticoagulant treatment period
* Patients with a current overt bleeding or known haemorrhage condition (e.g. active G.I. ulcer)
* Patients with a platelet count < 100 x 10 9/L
* Patients with a known history of heparin-induced thrombocytopenia
* Patients with known severe hepatic insufficiency manifested as international normalized ratio (INR) greater than or equal to 1.5
* Patients with uncontrolled severe hypertension i.e. a systolic blood pressure > 220 mm Hg or diastolic blood pressure > 120 mm Hg during at least 2 measurements within 24 hours prior to randomisation
* Patients with ischaemic stroke at or within last 1 week prior to randomisation
* Patients with a known haemorrhagic stroke within 3 months prior to randomisation
* Patients with known bacterial endocarditis within 3 months prior to randomisation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 541 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Leizorovicz, MD, Principal Investigator — Faculté de Médecine Laënnec
Locations (9):
- Bulgaria - managed by CRO, Sofia, Bulgaria
- Croatia - managed by CRO, Zagreb, Croatia
- Czech Republic - managed by CRO, Prague, Czechia
- Hôpital de la Cavale Blanche, Brest, France
- Med. Klinik IV/Klinikum Darmstadt, Darmstadt, Germany
- Klinika Chirugii Naczyniowej, Szczecin, Poland
- Romania - managed by CRO, Bucharest, Romania
- Clinical Center Serbia, Institute of Cardiovascular diseases & Centre for Vascular Surgery-Belgrade, Belgrade, Serbia
- Service of Geriatry, Hospital Universitario Clínico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leizorovicz A, Siguret V, Mottier D; Innohep(R) in Renal Insufficiency Study Steering Committee; Leizorovicz A, Siguret V, Mottier D, Clonier F, Janas M, Stinson J, Townshend G, Maddalena M. Safety profile of tinzaparin versus subcutaneous unfractionated heparin in elderly patients with impaired renal function treated for acute deep vein thrombosis: the Innohep(R) in Renal Insufficiency Study (IRIS). Thromb Res. 2011 Jul;128(1):27-34. doi: 10.1016/j.thromres.2011.03.002. Epub 2011 Apr 7. PMID 21477846
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between Dec 2005 and May 2008
Pre-assignment Details: 2 patients were not randomized
Period: Overall Study
Arm/Group | Innohep® | Heparin
Started | 269 | 270
Completed | 232 | 246
Not Completed | 37 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Innohep® | Heparin | Total
Number analyzed (Participants) | 269 | 270 | 539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 269 | 270 | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.9 (5.7) | 82.6 (5.8) | 82.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 168 | 345
  Male | 92 | 102 | 194
Region of Enrollment [Number; unit: participants]
  Serbia | 37 | 43 | 80
  France | 139 | 139 | 278
  Poland | 0 | 1 | 1
  Spain | 39 | 38 | 77
  Romania | 30 | 20 | 50
  Croatia | 9 | 16 | 25
  Germany | 10 | 10 | 20
  Belgium | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinically Relevant Bleeding Events
Time Frame: prior to day 90 +/- 5
Population: 2 patients randomised to the Heparin group withdrew their consent just after randomisation and before taking any study treatment. No data were collected after visit 1, and due to the nature of the withdrawal, no further information was possible to collect. These patients were excluded from all analyses
Measure: Number; unit: Patients
Arm/Group | Innohep® | Heparin
Number analyzed (Participants) | 269 | 268
Patients | 32 | 32

2. Secondary Outcome: Number of Patients With Recurrence of Venous Thromboembolism
Time Frame: prior to day 90 +/- 5
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Innohep® | Heparin
Number analyzed (Participants) | 269 | 268
Patients | 16 | 9

3. Secondary Outcome: Number of Patients With Major Bleeding Events
Time Frame: prior to day 90 +/- 5
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Innohep® | Heparin
Number analyzed (Participants) | 269 | 268
Patients | 12 | 10

ADVERSE EVENTS:
Description: Five patients who did not receive any study treatment were excluded from the safety analysis set. Three patients randomised to the Heparin group received innohe® during all their SC treatment period by mistake. These three patients were accounted for with respect to the trial medication actually taken, i.e. innohep®, in the safety analysis set.
Arm/Group | Innohep® | Heparin
Serious Adverse Events (participants affected / at risk) | 63/270 | 52/264
Other Adverse Events (participants affected / at risk) | 66/270 | 72/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Innohep® (N=270) | Heparin (N=264)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 6 | 6
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Thyrotoxicosis (Endocrine disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 2 | 2
Heparin-induced thrombocytopenia (General disorders) | 0 | 2
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 0
Sudden death (General disorders) | 2 | 2
Terminal state (General disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pneumonia escherichia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 4 | 2
Sepsis secondary (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Biopsy liver (Investigations) | 1 | 0
Coagulation time prolonged (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 1
International normalised ratio increased (Investigations) | 2 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Sigmoidoscopy (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis acquired (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dependence on respirator (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Amputation (Surgical and medical procedures) | 1 | 0
Anticoagulant therapy (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Pneumatic compression therapy (Surgical and medical procedures) | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 2
Embolism (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 5 | 3
Ischaemia (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebothrombosis (Vascular disorders) | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Innohep® (N=270) | Heparin (N=264)
Constipation (Gastrointestinal disorders) | 17 | 23
Diarrhoea (Gastrointestinal disorders) | 12 | 15
Urinary tract infection (Infections and infestations) | 25 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 14
Haematoma (Vascular disorders) | 21 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less